CLINICAL TRIAL: NCT01921673
Title: A Phase I-II Trial of Dovitinib Plus Docetaxel as Second-line Chemotherapy in Patients With Metastatic or Unresectable Gastric Cancer After Failure of First-line Chemotherapy
Brief Title: Dovitinib Plus Docetaxel in Gastric Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Yoon-Koo Kang, Professor, Asan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMC1302
Record Dates: First submitted 2013-08-10; First posted 2013-08-13 (Estimated); Last update posted 2017-07-14 (Actual); Status verified 2017-07

CONDITIONS: Gastric Cancer
Keywords: Gastric cancer; Phase I/II; Second-line chemotherapy; Dovitinib; Docetaxel; Refractory to first-line chemotherapy
MeSH Terms: conditions — Stomach Neoplasms | interventions — 4-amino-5-fluoro-3-(5-(4-methylpiperazin-1-yl)-1H-benzimidazol-2-yl)quinolin-2(1H)-one; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dovitinib plus docetaxel (Experimental): In phase I portion of the study Docetaxel 45-75 mg/m2, intravenous, every 3 weeks Dovitinib 200-500 mg, oral, 5 days on/2 days off
  In phase II portion of the study Recommended dose of docetaxel and dovitinib in phase I portion will be used.
  Interventions: Drug: Dovitinib and docetaxel

INTERVENTIONS:
Drug: Dovitinib and docetaxel — In phase I portion of the study Docetaxel 45-75 mg/m2, intravenous, every 3 weeks Dovitinib 200-500 mg, oral, 5 days on/2 days off
  In phase II portion of the study Recommended dose of docetaxel and dovitinib in phase I portion will be used.

SUMMARY:
Docetaxel is currently one of standard second-line therapy in patients with gastric cancer. As angiogenesis and FGFR pathway has been suggested to be associated with gastric cancer, dovitinib, dual VEGFR and FGFR inhibitor, may have the potential to improve the outcomes of patients with gastric cancer. Therefore, we investigated the combination regimen of docetaxel and dovitinib.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically proven metastatic or unresectable adenocarcinoma of stomach or gastroesophageal junction
2. Patients with progressive disease (radiological confirmation required) after one line of chemotherapy except taxane for advanced gastric cancer in palliative setting
3. Presence of at least one evaluable disease by Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1
4. Age of 18 to 74 years
5. Estimated life expectancy of more than 3 months
6. Eastern Cooperative Oncology Group (ECOG) performance status 0~2
7. Adequate bone marrow function (Absolute neutrophil counts ≥ 1,500/uL, hemoglobin ≥ 8.0g/dL, and platelet ≥ 100,000/uL)
8. Adequate renal function (creatinine < 1.5mg/dL)
9. Adequate hepatic function (total bilirubin < 1.5 mg/dL, transaminase < 3 times the upper normal limit [5 times for patients with liver metastasis])
10. No prior anti-angiogenic therapy (anti-VEGF or VEGFR tyrosine kinase inhibitor etc) or FGF/FGFR inhibitor
11. No prior radiation therapy within 4 weeks of the study (Irradiated lesions should not be included in the evaluable lesions.)
12. Written informed consent

Exclusion Criteria:

1. Past or concurrent history of neoplasm other than gastric adenocarcinoma, except for curatively treated non-melanoma skin cancer or in situ carcinoma of the cervix uteri
2. Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to study treatment start
3. Bowel obstruction
4. Evidence of serious gastrointestinal bleeding
5. Presence of central nervous system (CNS) metastasis
6. History of significant neurologic or psychiatric disorders
7. Significant cardiac disease within 6 months of the study (congestive heart failure uncontrollable by medication, symptomatic coronary heart disease, or arrhythmia, myocardial infarction)
8. Left ventricular ejection fraction (LVEF) assessed by 2-D echocardiogram (ECHO) or multiple gated acquisition scan (MUGA), < 45%
9. Uncontrolled hypertension defined by a SBP ≥ 160 mm Hg and/or DBP ≥ 100 mm Hg, with or without anti-hypertensive medication. Initiation or adjustment of antihypertensive medication (s) is allowed prior to study entry.
10. QTc > 480 msec on screening ECG
11. Proteinuria defined by NCI CTCAE grade > 1 at baseline as measured by a urine dipstick (2+ or greater) and confirmed by a 24 hour urine collection ( > 1g/24hrs). Subjects may be re-screened if blood pressure is shown to be controlled with or without intervention
12. History of thrombotic or bleeding diathesis or coagulopathy
13. Serious non-healing wound, peptic ulcer, or bone fracture
14. Abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months
15. Pregnant or lactating women, women of childbearing potential not employing adequate contraception
16. Other serious illness or medical conditions

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2013-08 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose | 6 months
  If dose limiting toxicities are experienced in two or more out of six patients in the cohort (more than 33% of patient cohort), that dose will be defined as the maximum tolerated dose.
Progression-free survival | 2 year
  Progression-free survival is defined as the time from the first treatment to the onset of progressive disease or to the date of death whichever comes first.

SECONDARY OUTCOMES:
Response rate | 2 year
  Proportion of patients with complete and partial response according to the Response Evaluation Criteria in Solid Tumors version 1.1
Toxicity | 2 years
  Adverse events caused by study drugs according to the National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0
Overall survival | 2 years
  Time from start of study treatment to any cause of death
Biomarker | Baseline and 2 weeks after study treatment
  FGFR2 copy number will be evaluated in blood and tumor tissue. Treatment efficacy including overall response rate, progression-free survival, and overall survival will be compared according to FGFR2 copy number determined by both FISH and real time PCR using TaqMan probe.

CONTACTS AND LOCATIONS:
Overall Officials: Yoon-Koo Kang, M.D., Ph.D., Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea

REFERENCES:
- [Background] Lee JL, Ryu MH, Chang HM, Kim TW, Yook JH, Oh ST, Kim BS, Kim M, Chun YJ, Lee JS, Kang YK. A phase II study of docetaxel as salvage chemotherapy in advanced gastric cancer after failure of fluoropyrimidine and platinum combination chemotherapy. Cancer Chemother Pharmacol. 2008 Apr;61(4):631-7. doi: 10.1007/s00280-007-0516-6. Epub 2007 May 23. PMID 17520252
- [Background] Wesche J, Haglund K, Haugsten EM. Fibroblast growth factors and their receptors in cancer. Biochem J. 2011 Jul 15;437(2):199-213. doi: 10.1042/BJ20101603. PMID 21711248
- [Background] Yamamoto S, Yasui W, Kitadai Y, Yokozaki H, Haruma K, Kajiyama G, Tahara E. Expression of vascular endothelial growth factor in human gastric carcinomas. Pathol Int. 1998 Jul;48(7):499-506. doi: 10.1111/j.1440-1827.1998.tb03940.x. PMID 9701011